CLINICAL TRIAL: NCT05938933
Title: Personalized Health Planning--Shared Medical Appointments for Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 066.FAM.2019.C
Record Dates: First submitted 2021-12-09; First posted 2023-07-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Obesity
Keywords: personalized health planning; shared medical appointments
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Experimental): Cohort
  Interventions: Behavioral: PHP; Behavioral: SMA

INTERVENTIONS:
Behavioral: PHP — personalized health planning (PHP)
Behavioral: SMA — shared medical appointments (SMAs)

SUMMARY:
Obesity affects a large portion of our population and accounts for a significant individual health burden for both individual patients and society. Though as little as 3 to 5% weight loss is associated with significant clinical benefits,1,2 current approaches to treat patients with obesity are not providing patients with the interventions needed to routinely see this change. One potential solution to this problem is utilizing personalized health planning (PHP) shared medical appointments (SMAs) to address the treatment of obesity. As PHP SMA has shown to improve clinical outcomes and patient satisfaction when compared to traditional care in other chronic illnesses,3,4 it could also be useful as a strategy to improve the efficiency and effectiveness of treating patients with obesity.

DETAILED DESCRIPTION:
There will be 14 total participants in this study. All will be current patients enrolled at the Methodist Charlton Family Medicine Clinic in Dallas, TX. Female and male patients will be selected based on individual provider recommendations within the Family Medicine Clinic at Methodist Charlton Medical Center (Dallas, TX).

Obesity affects a large portion of our population and accounts for a significant individual health burden for both individual patients and society. Though as little as 3 to 5% weight loss is associated with significant clinical benefits,1,2 current approaches to treat patients with obesity are not providing patients with the interventions needed to routinely see this change. One potential solution to this problem is utilizing personalized health planning (PHP) shared medical appointments (SMAs) to address the treatment of obesity. As PHP SMA has shown to improve clinical outcomes and patient satisfaction when compared to traditional care in other chronic illnesses,3,4 it could also be useful as a strategy to improve the efficiency and effectiveness of treating patients with obesity. PHP tailors health care to the needs, values, and preferences of the individual patient. It facilitates the use of the best available resources for proactive, predictive medicine while recognizing the value of engaging patients in their care. Its clinical workflow allows for creation of a personal health plan for each patient in which shared patient-provider goals are outlined to address the patient's proximate and long-term health goals and risks.

The PHP model is flexible and adaptable to many clinical needs and settings. In the program described here, PHP is adapted for use within a SMA for individuals with obesity. SMAs are conducted in 90-minute group visits, wherein 8 to 12 patients meet together with a small clinical team that always includes a provider.

ELIGIBILITY:
Inclusion Criteria:

* Current patients enrolled at the Methodist Charlton Family Medicine Clinic in Dallas, TX.
* Female and male patients will be selected based on individual provider recommendations within the Family Medicine Clinic at Methodist Charlton Medical Center (Dallas, TX)
* Patients will include motivated adults in our clinic from the ages of 30 to 60 yrs old with BMI ranges of 35 to 50 without significant mood or cardio-pulmonary issues.
* If a patient does have diabetes mellitus (DM), it needs to be under reasonable control (i.e., A1C less than 9).

Exclusion Criteria:

* uncontrolled depression with a Patient Health Questionnaire-9(PHQ-9) score greater than 9
* history of bariatric surgery or future plans for bariatric surgery
* wheelchair bound
* uncontrolled chronic obstructive pulmonary disease (COPD)/asthma or supplemental oxygen dependence
* uncontrolled congestive heart failure (CHF)
* uncontrolled DM with A1C greater than 9
* pregnancy
* active cancer

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
weight change | within Seven Months
  tracked over the duration of the study for each participant and the effectiveness of the intervention will be determined by reductions in patients' post-intervention weight and percent weight loss.

SECONDARY OUTCOMES:
change in blood pressure | within seven months
  Blood pressure measures over the duration of the study
Change in waist circumferences | within seven months
  Measurement of waist circumferences over the period of study
Depression | within seven months
  depression will be measured by observation over the duration of the study
change in glycated hemoglobin percentage( A1C) | within seven months
  Different measures for A1C over the

CONTACTS AND LOCATIONS:
Overall Officials: Khadija Kabani, DO, Principal Investigator — Methodist Charlton Family Medicine
Locations (1):
- Methodist Charlton Family Medicine, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No